CLINICAL TRIAL: NCT02887586
Title: The Effectiveness and Mechanism Study of Auricular Needling in Treating Cancer Induced Anorexia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 81573958
Record Dates: First submitted 2016-08-16; First posted 2016-09-02 (Estimated); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2017-12

CONDITIONS: Anorexia Nervosa; Cancer
Keywords: Auricular Needling; Mechanism Study; Anorexia; Cancer
MeSH Terms: conditions — Anorexia Nervosa; Neoplasms; Anorexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Auricular Needling group (Experimental): Patients will receive auricular needling for 4 weeks .
  Interventions: Other: auricular needling
- control group (No Intervention): This group will receive no treatment. Subjects will be assessed at baseline and the 2th, 4th and 8th week.

INTERVENTIONS:
Other: auricular needling — Patients will be treated with auricular needling for 4 weeks. 4-8 specific auricular acupoints are selected unilaterally at a time, and alternate to another side every 2-3 days, treatment will last for 4 consecutive weeks. The following 4 ear acupoints points will be selected for every patient: Ear Shenmen, Stoma, Spleen, and Subcortex. Other ear acupoints including Triple Energizer, Liver, Sympathetic Nerve and Smallintestine will be selected based on the condition of patients. Treatment will be performed by a registered Chinese medicine practitioner.
  Arms: Auricular Needling group

SUMMARY:
Controlling of cancer induced anorexia is highly demanded by advanced cancer patients. It plays an important role in improving the quality of life among advanced cancer patients. Through a randomized controlled single blinded clinical research, we will observe the differences of appetite, food intake amount, weight and KPS between the auricular needling treating group and control group before and after the treatment. Based on the results of the research, we can prove the clinical effectiveness of auricular needling in treating cancer induced anorexia and possible mechanism of the method.

DETAILED DESCRIPTION:
Patients will be recruited from Xiyuan Hospital. In this study, eligible participants will be randomly assigned to two groups. In the auricular needling treating group, patients will receive needling treating for 4 weeks(auricular needles are given to one ear every time for 2-3days,then switch to the other). Conventional nutrition support and symptomatic treatment are given at the same time. In the control group, patient just receive conventional nutrition support and symptomatic treatment.

The simple appetite questionnaire, a symptom based Anorexia assessment questionnaire and fatigue symptom inventory questionnaire are used to assess the condition of patients. Other observation index include weight, KPS, appetite and the expectation of patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of malignant cancer of stage III or IV
* Meet the diagnosis criteria of cancer induced anorexia
* Karnofsky performance status(KPS) score≥ 60
* Expected survival time≥3 months
* Willing to give informed consent
* Able to comply with trial protocol

Exclusion Criteria:

* have blood routine, hepatic and renal disfunction,which is over 2 times of the normal value
* obvious eating disorder, intestinal obstruction, poor controlled heart disease and diabetes
* who are receiving progesterone, glucocorticoid or other hormone Therapy
* those who are participating in other trials.
* pregnant women, nursing mother or psychotic patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bin He, Principal Investigator — Xiyuan Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Xiyuan Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Auricular Needling Group: Patients will receive auricular needling for 4 weeks .
  auricular needling: Patients will be treated with auricular needling for 4 weeks. 4-8 specific auricular acupoints are selected unilaterally at a time, and alternate to another side every 2-3 days, treatment will last for 4 consecutive weeks. The following 4 ear acupoints points will be selected for every patient: Ear Shenmen, Stoma, Spleen, and Subcortex. Other ear acupoints including Triple Energizer, Liver, Sympathetic Nerve and Small intestine will be selected based on the condition of patients. Treatment will be performed by a registered Chinese medicine practitioner.
Period: Overall Study
Arm/Group | Auricular Needling Group | Control Group
Started | 30 | 30
Completed | 27 | 28
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Population: Fall off in 5 cases, fall off reason : active request exit in 1 case, disease progression can not complete treatment in 1 case, 3 cases of loss rate 8.3 %.
Groups:
- Total: Total of all reporting groups
Arm/Group | Auricular Needling Group | Control Group | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Categorical [Count of Participants; unit: Participants] — The mean age of these 55 participants was 65±11 (range, 31 to 80) years old.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 10 | 16 | 26
    >=65 years | 17 | 12 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] — The mean age of these 55 participants was 65±11 (range, 31 to 80) years old.
  years | 67 (7) | 63 (13) | 65 (11)
Sex: Female, Male [Count of Participants; unit: Participants] — 15 males and 13 females in control group and 10 males and 17 females in ear acupuncture group .
  Participants
    Female | 17 | 13 | 30
    Male | 10 | 15 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 27 | 28 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — All participants are from China.
  participants
    China | 27 | 28 | 55
Body weight [Mean (Standard Deviation); unit: kg] | 56.89 (10.04) | 58.47 (6.85) | 57.49 (8.55)

OUTCOME MEASURES:

1. Primary Outcome: Simple Appetite Questionnaire
Description: The Simplified Nutritional Appetite Questionnaire (SNAQ) is used to assess the patient's appetite.Possible scores range from 4（poor appetite) to20（good appetite）.The score lower than 14 predicts a risk of 5% weight loss.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Auricular Needling Group | Control Group
Number analyzed (Participants) | 27 | 28
score on a scale
  Baseline | 8.7 (1.996) | 9.57 (1.854)
  Treatment for 2 weeks | 11.26 (2.246) | 9.93 (1.654)
  Treatment for 4 weeks | 13.19 (2.058) | 9.50 (2.186)
  Stop treatment for 4 weeks | 13.00 (2.236) | 9.68 (2.161)

2. Primary Outcome: Symptom Based Anorexia Assessment
Description: Symptom based anorexia assessment is used to evaluate whether and to what extent anorexia occurs in cancer patients.Possible scores range from 0(normal appetite) to 48(severe anorexia).After the patient answers all the questions in the table, the score is scored, and the final score is less than or equal to 24 points, which can be determined as anorexia.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Auricular Needling Group | Control Group
Number analyzed (Participants) | 27 | 28
score on a scale
  Baseline | 8.70 (1.996) | 9.57 (1.854)
  Treatment for 2 weeks | 11.26 (2.246) | 9.93 (1.654)
  Treatment for 4 weeks | 13.19 (2.058) | 9.5 (2.186)
  Stop treatment for 4 weeks | 13.00 (2.236) | 9.68 (2.161)

3. Secondary Outcome: Appetite Improvement
Description: The appetite improvement is used to indicates the patient's appetite.Method: Use a moving ruler about 10cm long, with one side marked with 10 scales, the two ends are "0" and "10" respectively, 0 means normal appetite, 10 scores indicate extreme aversion to food. When in use, the side with the scale should face away from the patient, and let the patient mark on the ruler.The corresponding position that can represent one's own desire for food, the position marked by the doctor according to the patient is its score, clinical evaluation is divided into "normal appetite/basically normal eaters", "3-5" with "0-2".
  Divided into "mild anorexia", "6-8" into "moderate anorexia", >8 into "severe anorexia"
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Auricular Needling Group | Control Group
Number analyzed (Participants) | 27 | 28
score on a scale
  Baseline | 6.56 (1.717) | 5.39 (1.548)
  Treatment for 2 weeks | 4.56 (2.172) | 5.36 (1.496)
  Treatment for 4 weeks | 3.59 (1.845) | 5.29 (1.823)
  Stop treatment for 4 weeks | 3.30 (1.918) | 5.75 (1.818)

4. Secondary Outcome: Weight
Description: Weight used to assess the appetite of patient.Body weight changes caused by factors such as body cavity effusion and edema were excluded. Improvement: weight gain > 2kg,and maintained for more than 4 weeks. Stable: Weight gain or loss ≤ 2kg. Exacerbation: Weight loss > 2kg.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Auricular Needling Group | Control Group
Number analyzed (Participants) | 27 | 28
kg
  Baseline | 56.89 (10.040) | 58.47 (6.851)
  Treatment for 2 weeks | 57.32 (9.741) | 58.30 (6.922)
  Treatment for 4 weeks | 58.05 (9.998) | 57.86 (6.751)
  Stop treatment for 4 weeks | 58.08 (9.753) | 57.54 (6.964)

5. Secondary Outcome: Acupuncture Treating Expectation Questionnaire
Description: Acupuncture treating expectation questionnaire used to assess patients' expectation for auricular needling.Higher scores indicate higher expectations.Possible scores range from 4（low expectations） to 20（high expectations).
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Auricular Needling Group | Control Group
Number analyzed (Participants) | 27 | 28
score on a scale
  baseline | 12.26 (3.68) | 10.00 (4.42)
  Treatment for 2 weeks | 13.74 (3.25) | 9.64 (3.73)
  Treatment for 4 weeks | 14.30 (3.30) | 9.04 (4.38)
  Stop treatment for 4 weeks | 11.04 (5.09) | 7.57 (4.02)

ADVERSE EVENTS:
Time Frame: ten weeks.
Arm/Group | Auricular Needling Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-05-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT02887586/Prot_000.pdf
  • Statistical Analysis Plan (2016-05-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT02887586/SAP_001.pdf
  • Informed Consent Form (2016-05-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT02887586/ICF_002.pdf